CLINICAL TRIAL: NCT00226330
Title: A Double-Blind, Multi-Centre, Active-Controlled (15, 30, and 45 mg Pioglitazone) Long-Term Extension Study to Evaluate the Safety and Tolerability of Tesaglitazar (0.5 and 1 mg) in Patients With Type 2 Diabetes Mellitus (GALLEX 6)
Brief Title: GALLEX 6: Study to Evaluate the Safety and Tolerability of Tesaglitazar in Patients With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The development program has been terminated
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6160C00048
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Patients diagnosed with type 2 diabetes who have participated in and completed the randomized, double-blind, parallel-group, multi-center study GALLANT 6.
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tesaglitazar; Pioglitazone

INTERVENTIONS:
Drug: Tesaglitazar — (0.5 or 1 mg)
  Other Names: Galida
Drug: Pioglitazone — (15, 30 or 45 mg)
  Other Names: Actos

SUMMARY:
This is a parallel-group, multi-center, long-term extension study from the GALLANT 6 study to monitor the safety and tolerability of oral tesaglitazar compared with pioglitazone in patients with type 2 diabetes for up to 104 weeks of treatment. The total duration, including treatment and follow-up, is 107 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Men or women who are >= 18 years of age
* Female patients: postmenopausal; hysterectomized; or, if of childbearing potential, using a reliable method of birth control.
* Completed the last two visits of the randomized treatment period in GALLANT 6

Exclusion Criteria:

* Type 1 diabetes
* New York Heart Association heart failure Class III or IV
* Treatment with chronic insulin
* History of hypersensitivity or intolerance to any peroxisome proliferator-activated receptor agonist (like Actos or Avandia), fenofibrate, metformin or 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor (statin)
* History of drug-induced myopathy or drug-induced creatine kinase elevation, liver enzyme elevations, or neutropenia (low white blood cells)
* Creatinine levels of above twice the normal range
* Creatine kinase of above 3 times the upper limit of normal
* Previous enrollment in this long-term extension study
* Any clinically significant abnormality identified by physical examination, laboratory tests or electrocardiogram, which, in the judgment of the investigator, would compromise the patient's safety or successful participation in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100
Dates: Start 2005-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Adverse events
Laboratory variables
Physical examination
Cardiac evaluation
Hypoglycemic events
Electrocardiogram
Vital signs (blood pressure and pulse)
Body weight

SECONDARY OUTCOMES:
Pharmacodynamic: fasting plasma glucose, glycosylated hemoglobin A1c
Lipid variables (triglyceride, total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol [HDL-C], and non-HDL-C)
Responder rates and proportion of patients on tesaglitazar who reach pre-specified target levels for triglyceride, total cholesterol, low-density lipoprotein cholesterol, HDL-C and non-HDL-C
C-reactive protein (CRP)
Central obesity (waist circumference, hip circumference, waist/hip ratio)
Patient reported outcomes using the Medical Outcomes Study Short Form-36 (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Galida Medical Science Director, MD, Study Director — AstraZeneca
Locations (171):
- United States (110):
  - Research Site, Birmingham, Alabama
  - Research Site, Columbiana, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Sierra Vista, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Searcy, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Carmichael, California
  - Research Site, Dinuba, California
  - Research Site, Elk Grove, California
  - Research Site, Encinitas, California
  - Research Site, Encino, California
  - Research Site, Fresno, California
  - Research Site, Greenbrae, California
  - Research Site, Loma Linda, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Northridge, California
  - Research Site, Pasadena, California
  - Research Site, Redondo Beach, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, Santa Ana, California
  - Research Site, Santa Monica, California
  - Research Site, Spring Valley, California
  - Research Site, Tustin, California
  - Research Site, Walnut Creek, California
  - Research Site, West Hills, California
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Brandon, Florida
  - Research Site, Cooper City, Florida
  - Research Site, Delray Beach, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocoee, Florida
  - Research Site, Orlando, Florida
  - Research Site, Plantation, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Dunwoody, Georgia
  - Research Site, Berwyn, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Elk Grove Village, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Melrose Park, Illinois
  - Research Site, North Chicago, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Sterling, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Waterloo, Iowa
  - Research Site, Topeka, Kansas
  - Research Site, Witchita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Haverhill, Massachusetts
  - Research Site, Petoskey, Michigan
  - Research Site, Excelsior Springs, Missouri
  - Research Site, Richmond Heights, Missouri
  - Research Site, Rolla, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, North Las Vegas, Nevada
  - Research Site, Pahrump, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Pleasantville, New Jersey
  - Research Site, Manlius, New York
  - Research Site, New York, New York
  - Research Site, Olean, New York
  - Research Site, Staten Island, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Lakewood, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Reading, Pennsylvania
  - Research Site, Warminster, Pennsylvania
  - Research Site, West Chester, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Carrollton, Texas
  - Research Site, Dallas, Texas
  - Research Site, North Richland Hills, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Norfolk, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Gig Harbor, Washington
  - Research Site, Huntington, West Virginia
- Argentina (6):
  - Research Site, Morón, Buenos Aires
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba - Córdoba
  - Research Site, Rosario
  - Research Site, Salta - Salta
- Brazil (6):
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, São Paulo
- Canada (22):
  - Research Site, Edmonton, Alberta
  - Research Site, Abbotsford, British Columbia
  - Research Site, Chilliwack, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Dartmouth, Nova Scotia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Truro, Nova Scotia
  - Research Site, Windsor, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Niagara Falls, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, St. Catharines, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Trois-Rivières, Quebec
- Finland (6):
  - Research Site, Helsinki
  - Research Site, Jakobstad
  - Research Site, Kauniainen
  - Research Site, Kuopio
  - Research Site, Pori
  - Research Site, Tampere
- Mexico (6):
  - Research Site, Guadalajara, Jalisco.
  - Research Site, México, D.F.
  - Research Site, Nuevo León, Monterrey
  - Research Site, Puebla, Mexico
  - Research Site, Torreón
  - Research Site, Zapopan
- United Kingdom (15):
  - Research Site, Belfast
  - Research Site, Cardiff
  - Research Site, Co Antrim N Ireland
  - Research Site, Co. Wexford, Ireland
  - Research Site, Dublin
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Kent
  - Research Site, Leeds
  - Research Site, Mid Glamorgan
  - Research Site, Pembrokeshire
  - Research Site, Plymouth
  - Research Site, Reading
  - Research Site, Surrey
  - Research Site, Wiltshire